CLINICAL TRIAL: NCT05360862
Title: Effects of Prone Positioning-induced on the Recruitment-to-inflation Ratio in COVID-19 Patients With Acute Respiratory Distress Syndrome
Brief Title: Prone Positioning and R/I Ratio in COVID-19 Patients With ARDS (SyDRAC-DV)
Acronym: SyDRAC-DV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22-PP-02
Record Dates: First submitted 2022-05-03; First posted 2022-05-04 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: ARDS; COVID-19; Prone positioning; Lung recruitement
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prone positioning session
  Interventions: Procedure: Prone positioning session

INTERVENTIONS:
Procedure: Prone positioning session — To perform respiratory measurements before, during and after a prone positioning session.

SUMMARY:
The purpose of this study is to determine the efects of prone positioning on the recruitment- to-inflation ratio in COVID-19 patients with acute respiratory distress syndrome.

DETAILED DESCRIPTION:
High positive end-expiratory pressure (PEEP) level and prone positioning (PP) are recommended in patients with moderate to severe acute respiratory distress syndrome (ARDS) in order to recruit lung and thus to improve oxygenation. Thus, high PEEP level and prone positioning will be more effective in patients with high potential for lung recruitment. Recently, the Recruitment-to-Inflation Ratio (R/I ratio) has been described and validated in patients with ARDS to estimate the potential for lung recruitment. In this regard, the R/I ration may be of interest to titrate PEEP level in patients with ARDS. This would be of particular interest in COVID-19 patients with ARDS, since different ARDS phenotypes with heterogeneous potential of lung recruitment have been described in these patients. However, the effects of prone positioning on R/I ratio have been scarcely described so far. Thus, the main goal of this study is to investigate the effects of prone positioning on the R/I ratio in COVID-19 patients with ARDS. The second goal of this study is to determine the effects of prone positioning on oxygenation and respiratory mechanics according to the R/I ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive mechanical ventilation
2. Patients with acute respiratory distress syndrome according to the Berlin definition
3. Positive COVID-19 real-time reverse transcriptase-polymerase chain reaction assay in nasal swabs or pulmonary samples.
4. Indication to a prone positioning session by the attending physician

Exclusion Criteria:

1. Age <18 years and pregnant women
2. Patients under legal protection
3. Acute core pulmonale
4. Pneumothorax and/or chest drainage
5. Hemodynamic failure

   1. Increase in norepinephrine dosage >30% within the last 6 hours
   2. Norepinephrine dosage > 0.5 mg/kg/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are COVID-19 patients with moderate to severe ARDS under mechanical ventilation in whom prone positioning is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Prone positioning-induced decrease in R/I ratio. | 16-hour prone positioning session and 4-hour period after supine repositioning
  The R/I ratio will be calculated before (within 30 minutes before), during (2h, 8h and 16h) and after (2h and 4h after) a prone positioning session.

SECONDARY OUTCOMES:
Proportion of patients "responders" to prone positioning session | 16-hour prone positioning session and 4-hour period after supine repositioning
  The R/I ratio will be calculated before (within 30 minutes before), during (2h, 8h and 16h) and after (2h and 4h after) a prone positioning session.
Clinical and respiratory predictors of prone positioning response in terms of oxygenation | 16-hour prone positioning session and 4-hour period after supine repositioning
  TROC curves of clinical and biological variables for prediction of response to prone positioning

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
No sharing data plan is sheduled.